### INFORMED CONSENT FORM

#### Informed Consent form

# TITLE: Process evaluation of the effectiveness of two transdiagnostic interventions targeting emotional regulation: compassion focused program and emotional skills training program

| N°ID RCB | N°CPP | N°CNIL |
|----------------|-----------------|---------|
| 2020-A00551-38 | 2020.09.03 ter_ | 2217007 |
| | 20.05.13.42837 | |

Document date: 17/01/2021

**Study sponsor and investigator**: **Mathias Butaud,** Psychiatrist 4 avenue Jean Perrot, 38000 Grenoble

**Co-investigator** : **Céline Baeyens**, Professor, Laboratoire Inter-universitaire de Psychologie, Université Grenoble Alpes, UFR SHS, 1251 avenue Centrale, CS 40700, 38058 Grenoble Cedex 9

Associated investigators: Rebecca Bègue-Shankland, Professor au Laboratoire Développement, Individu, Processus, Handicap, Education (DIPHE), Université Lyon 2, Bâtiment V (V211 à V216), 5, Avenue Pierre Mendès-France, 69676 Bron Cedex, Marine Paucsik, PhD STudent, Laboratoire Interuniversitaire de Psychologie, Université Grenoble Alpes, UFR SHS, 1251 avenue Centrale, CS 40700, 38058 Grenoble Cedex 9, Francis Gheysen, psychiatrist, 1 avenue du 6 juin, 14000 Caen, Benjamin Gouache, psychiatrist, Claire Cécile Périer et Rocio Roure, neuropsychologist – Centre Référent de Réhabilitation Psychosociale et de Remédiation cognitive (C3R) de Grenoble, Centre Ambulatoire de Santé Mentale, 8 place du Conseil de la Résistance, 38100 Saint-Martin-d'Hères, Laure Favre-Réguillon, Psychologist – Centre Référent de Réhabilitation Psychosociale et de Remédiation cognitive (C3R) de Grenoble, Centre Ambulatoire de Santé Mentale, 8 place du Conseil de la Résistance, 38100 Saint-Martin-d'Hères, Céline Roussel, psychiatrist et Sandrine Rebelle, neuropsychologist, Centre départemental de réhabilitation psychosociale des Glières 219, Chemin des bois des Fornets 74800 La Roche-sur-Foron.

## **Participant**

| l, | , declare that I have been informed about the nature of |
|---|---|
| the study | , its purpose, duration, possible benefits and risks and what is expected of me. I have |
| read the | information document and the appendix to this document. |

I have had enough time to think about it and talk about it with someone I choose, such as my doctor or a family member.

I had the opportunity to ask any questions that came to mind and my questions were answered to my satisfaction.

I understand that my participation in this study is voluntary and that I am free to end my participation in this study without affecting my relationship with the therapeutic team in charge of my health.

I understand that when I read and sign this consent form, I can be assisted by a trusted person as mentioned in article L.1111-6 CSP stipulating: "If the patient wishes, the trusted person

## INFORMED CONSENT FORM

accompanies him/her in his/her steps and attends medical interviews in order to help him/her in his/her decisions.

I understand that data about me will be collected during my participation in this study and that the investigating physician and the study sponsor guarantee the confidentiality of this data.

I consent to the processing of my personal data.

I agree that the research data collected for the purposes of this study may be further processed, provided that this processing is limited to the context of this study for the purpose of gaining a better scientific understanding of the effectiveness of psychotherapy.

I have received a copy of the participant information and informed consent.

| Name, first name, date and signature of the participant. |
|---|
| Investigating Doctor: |
| I, associate investigating doctor, confirm that I have provided the necessary information about the study and have provided a copy of the participant information document. |
| I confirm that no pressure has been exerted on the patient to agree to participate in the study and that I am prepared to answer any additional questions, if necessary. I confirm that I am working in accordance with the ethical principles set out in the latest version of the "Declaration of Helsinki", the "Good Clinical Practice" and the law of 7 May |
| 2004, relating to experiments on the human person. |
| Name, first name, date and signature of the associated investigator |